CLINICAL TRIAL: NCT03968055
Title: The Use of Continuous Glucose Monitor Technology and Remote Monitoring to Change Clinical Outcomes Following New Diagnosis of Type 1 Diabetes in the Pediatric Population
Brief Title: Remote Monitoring of CGM Data in Pediatric Patients With Newly Diagnosed Type 1 Diabetes (T1D)
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Priya Prahalad, Clinical Assistant Professor, Stanford University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 48935
Record Dates: First submitted 2019-05-28; First posted 2019-05-30 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Type 1 Diabetes
Keywords: pediatrics
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with Type 1 Diabetes (Other): Participants will wear a continuous glucose monitor (CGM) and receive remote monitoring of the CGM data by the clinical care team.
  Interventions: Other: Integration with Epic

INTERVENTIONS:
Other: Integration with Epic — Participants will have CGM data connected to our medical record through an already established pathway (Dexcom app on iOS device to Apple HealthKit to Epic MyChart to Epic)
  Other Names: GluVue Platform

SUMMARY:
To determine if increased targeted contact between patients and the care team can improve diabetes outcomes in the 1st year after diagnosis. We will be using the GluVue platform to remotely view continuous glucose monitor (CGM) data.

DETAILED DESCRIPTION:
Based on alerts from GluVue, care team members will proactively reach out to patients and their families for more frequent dose adjustments. We will assess if remote monitoring facilitates contact between the care team and patients and improves glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* All individuals within one month of T1D diagnosis seen at the Stanford Children's Diabetes Clinic
* Individuals who plan to receive follow up care at the Stanford Children's Diabetes Clinic
* Individuals who agree to CGM data integration into the electronic medical record (EMR) for remote monitoring
* Age: birth to < 21 years of age

Exclusion Criteria:

* Diabetes diagnosis other than T1D
* Diagnosis of diabetes > 1 month prior to initial visit
* Individuals with the intention of obtaining diabetes care at another clinic
* Individuals who do not consent to CGM use, CGM data integration, or remote monitoring
* Individuals > 21 years of age

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-03-25 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Contacts with the care provider | 1 year
  Prospective chart review to determine the number of contacts between the participant and care team due to remote monitoring

SECONDARY OUTCOMES:
Hemoglobin A1c | 1 year
  Prospective chart review for lab values

CONTACTS AND LOCATIONS:
Overall Officials: Priya Prahalad, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Prahalad P, Ding VY, Zaharieva DP, Addala A, Johari R, Scheinker D, Desai M, Hood K, Maahs DM. Teamwork, Targets, Technology, and Tight Control in Newly Diagnosed Type 1 Diabetes: the Pilot 4T Study. J Clin Endocrinol Metab. 2022 Mar 24;107(4):998-1008. doi: 10.1210/clinem/dgab859. PMID 34850024